CLINICAL TRIAL: NCT04926116
Title: A Phase I Study to Evaluate The Safety, Tolerability, and Pharmacokinetics of AK3280 in Chinese Healthy Volunteers
Brief Title: A Study of AK3280 in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK3280-2001
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AK3280 Cohort 1 (Experimental): Eligible subjects will be administered a single oral dose of 200 mg AK3280 under fasted conditions on Day 1. A multiple dosing period follows with daily 200 mg AK3280 b.i.d. administered with a concurrent low-fat meal intake from Day 4 to Day 16 and a 200 mg AK3280 q.d. dosing on Day 17.
  Interventions: Drug: AK3280
- AK3280 Cohort 2 (Experimental): The dose level of AK3280 for Cohort 2 will be determined by the SRC (Safety Review Committee) based on the safety and PK data gleaned in Cohort 1. Subjects will receive AK3280 following the same dosing schedule as that in Cohort 1, i. e., a single oral dose of AK3280 under fasted conditions on Day 1, multiple AK3280 b.i.d. administration with a concurrent low-fat meal intake from Day 4 to Day 16, and an AK3280 q.d. dose on Day 17.
  Interventions: Drug: AK3280
- AK3280 Optional Cohort (Experimental): This is an optional dose cohort that the SRC will determine depending on the results of Cohorts 1 and 2, including the proposed dose level. Potential subjects in this cohort will also follow the same dosing scheme as those for Cohorts 1 and 2.
  Interventions: Drug: AK3280
- Control Arm (Placebo Comparator): There are placebo controls in each dose cohort to assess the safety profile of the study medication. Subjects will be randomized to receive a placebo simultaneously as those subjects randomized to AK3280.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK3280 — Active Substance: AK3280, Pharmaceutical Form: Tablet, Route of Administration: Oral
  Arms: AK3280 Cohort 1; AK3280 Cohort 2; AK3280 Optional Cohort
Drug: Placebo — Active Substance: Placebo, Pharmaceutical Form: Tablet, Route of Administration: Oral
  Arms: Control Arm

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, single-center, phase I study to evaluate the safety, tolerability, and pharmacokinetics of AK3280 in healthy Chinese subjects.

DETAILED DESCRIPTION:
This phase I study is a randomized, double-blind, placebo-controlled, single-center clinical study in healthy subjects. The objectives of the study are to evaluate the safety, tolerability, and pharmacokinetics of AK3280. Approximately, 36 healthy Chinese subjects will be recruited and randomized to orally receive AK3280 or matching placebo. The total duration of the study will be approximately 25 days for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are willing to sign and date informed consent forms.
* Male or female participants between 18 and 45 years of age, inclusive.
* Have a bodyweight ≥50.0 kg (Male) or ≥45.0 kg (Female), and a body mass index (BMI) between 19.0 and 28.0 kg/m^2, inclusive.
* Participants are in good health without any significant clinical abnormalities on the basis of medical history related to heart, liver, kidneys, gastrointestinal tracts, or mental, central nervous, and metabolic disorders; physical examination (including vital signs); baseline laboratory test and 12-lead electrocardiogram (ECG) results.
* Participants (including male participants) who have no pregnancy plan and are willing to use an effective method of contraception during the screening period and for three months thereafter without sperm or egg donation plans.
* Participants who are capable to communicate with investigators and comply with the study requirements.

Exclusion Criteria:

* Allergic to any of the study drug ingredients or ineligible determined by the investigator due to a history of food or drug allergies.
* Having an abnormal medical history in terms of clinically significant digestive, urological, neurological, hematological, endocrine, oncological, pulmonary, immunological, cardiovascular, or psychiatric diseases or having histories of use any prescription, over-the-counter, herbs, vitamins, or vaccines within four weeks prior to study drug administration.
* Intolerant to venipuncture or having difficulty in venous blood collection.
* Having a personal history of drug and alcohol abuse, use of nicotine-containing products, receiving caffeine-containing drinks, taking grapefruit or food made of it, and medications, food, or beverages such as xanthines that could affect the ADME of study medication.
* Having clinically significant abnormalities in vital sign measures and lab test results.
* Female subjects are lactating at screening.
* Previous participation in any clinical trial within 3 months prior to screening.
* Inability to meet the study requirements in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects with Adverse Events (AEs) | From baseline up to approximately 6 weeks
  An adverse event can be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study medication, whether or not considered related to the study medication in this clinical trial.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of AK3280 | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The maximum observed plasma concentration of AK3280.
Maximum Observed Plasma Concentration (Cmax) of AK3280 Metabolite | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The maximum observed plasma concentration of AK3280 metabolite.
Observed trough plasma concentration at end of dosing interval (Ctrough) of AK3280 | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The concentration of AK3280 reached immediately before the next dose administered.
Observed trough plasma concentration at end of dosing interval (Ctrough) of AK3280 Metabolite | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The concentration of AK3280 metabolite reached immediately before the next dose administered.
Measure maximum plasma concentration at steady state (Css max) of AK3280 | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The maximum concentration of AK3280 reached at steady state.
Measure maximum plasma concentration at steady state (Css max) of AK3280 Metabolite | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The maximum concentration of AK3280 metabolite reached at steady state.
Time to Maximum Plasma Concentration (Tmax) of AK3280 | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The time of occurrence of Cmax of AK3280
Time to Maximum Plasma Concentration (Tmax) of AK3280 Metabolite | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The time of occurrence of Cmax of AK3280 metabolite
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) of AK3280 | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The area under the plasma concentration-time curve from time zero up extrapolated to infinity of AK3280.
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) of AK3280 Metabolite | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The area under the plasma concentration-time curve from time zero up extrapolated to infinity of AK3280 metabolite.
Area under the plasma concentration-time curve from time zero up to 12hrs (AUC 0-12h) of AK3280 | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8, and 12hours post-dose)
  The area under the plasma concentration-time curve from time zero up to the 12hrs analytically quantifiable concentration of AK3280.
Area under the plasma concentration-time curve from time zero up to 12hrs (AUC 0-12h) of AK3280 Metabolite | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8, and 12hours post-dose)
  The area under the plasma concentration-time curve from time zero up to the 12hrs analytically quantifiable concentration of AK3280 metabolite.
Terminal Half-Life (t1/2) of AK3280 | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The apparent elimination half-life of AK3280.
Terminal Half-Life (t1/2) of AK3280 Metabolite | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The apparent elimination half-life of AK3280 metabolite.
Apparent Oral Clearance (CL/F) of AK3280 | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The oral clearance of AK3280.
Apparent Oral Clearance (CL/F) of AK3280 Metabolite | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The oral clearance of AK3280 metabolite.
Apparent volume of distribution during terminal phase (Vz/F) of AK3280 | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The Vz/F of AK3280 will be calculated as CL/λz.
Apparent volume of distribution during terminal phase (Vz/F) of AK3280 Metabolite | Day1/Day17(pre-dose and 0.5,1,1.5,2,2.5,3,4,6,8,12hours post-dose), Day2/Day18(24hours post-dose), Day3/Day19(48hours post-dose), Day4/Day20(72hours post-dose); and Days6,8,10,14,15,16 (pre-dose)
  The Vz/F of AK3280 metabolite will be calculated as CL/λz.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Gu, Study Director — info@arkbiosciences.com
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No